CLINICAL TRIAL: NCT02099500
Title: An Open-label, Non-Randomized, Patient Funded, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Via Intramuscular Injections for the Treatment of Critical Limb Ischemia
Brief Title: Autologous Adipose-Derived Stromal Cell Delivered Via Intramuscular Injections for the Treatment of Critical Limb Ischemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-US-CLIN-001
Record Dates: First submitted 2014-03-19; First posted 2014-03-31 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Critical Limb Ischemia
Keywords: Critical Limb Ischemia; Peripheral Vascular Disease; Lower Limb Ulcer; Gangrene; Amputation; Lower Limb Wound
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases; Leg Ulcer; Gangrene | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell Injection (Experimental): Non-Randomized
  Interventions: Procedure: Liposuction; Other: Stem Cell Injection

INTERVENTIONS:
Procedure: Liposuction — Liposuction using aspiration syringe and tumescent local anesthesia
  Other Names: Adipose-Derived Stem Cells
Other: Stem Cell Injection — Stem cell implantation will be performed using intramuscular injection into the affected ischemic site of interest

SUMMARY:
This is an open-label, non-randomized, multi center, patient sponsored study of Adipose-Derived Stromal Cell (ASC) implantation via intramuscular injections in patients who have critical limb ischemia not amenable for revascularization.

The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the disease pathology of patients with diagnosed critical limb ischemia ASCs will be collected from the patient's adipose-derived tissue (body fat). Using local anesthesia, Liposuction will be performed to collect the adipose tissue specimen. The adipose tissue is then transferred to the laboratory for separation of the adipose tissue derived stem cells. In addition, peripheral blood will be collected for isolation of platelet rich plasma, which are then combined with the ASC's for intramuscular injection into the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* Age ~ 18 years
* Existence of limb ischemia, with clinical presentation corresponding to Rutherford Categories 2-6 as defined in the reporting standards adopted by \ the Society of Vascular Surgeons, or corresponding to the Leriche-Fontaine Classification, stages II, III, or IV
* Patients with, ischemia and ischemic ulceration provided patient have angiographic evidence of vascular compromise and is not a candidate for revascularization
* Stable and on optimal medical management for > 60 days as follows:
* Clopidogrel/aspirin therapy or other anticoagulation therapy, cholesterol- lowering agent, and⁄or antihypertensive medication
* Hematocrit ≥ 28.0%, White Blood Cell count ≤14,000, Platelet count ≥ 50,000
* Creatinine ≤ 2.5 mg/dL, and INR ≤ 1.6 (unless taking warfarin) or PTT < 1.5× control (to avoid bleeding complications). INR values for patients taking warfarin will be corrected prior to the procedure
* Patient meets at least one of the following diagnostic criteria for the index limb:

  1. ABI<.5mmHg
  2. TcpO2 <20 mm Hg when lying down and breathing room air, if available
  3. Or, nonhealing ulcer due to local arterial compromise with no opportunity for revascularization
* At least one non-healing distal extremity ischemic ulcer as confirmed by a vascular surgeon
* Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria:

* Female who is pregnant or nursing, or is of childbearing potential and not using a reliable method of contraception
* Any medical problems contraindicating tumescent syringe liposuction
* Life expectancy < 6 months
* Patient determined to be nonsurgical candidate due to reasons such as

  1. High-risk medical conditions
  2. Unstable cardiac disease
  3. Stroke or transient ischemic attack leading to limitations in lower extremities or occurring within 180 days prior to the initial screening visit
  4. Severe arthritis or other musculoskeletal disorder.
* Systolic blood pressure (supine) ≤ 90 mmHg
* Resting heart rate > 100 bpm
* Poorly controlled diabetes mellitus (HgbA1c > 10%)
* Life-threatening complications of limb ischemia necessitating immediate amputation
* Uncorrected iliac artery occlusion on index side unless corrected with stent
* Extensive necrosis of the index limb or other conditions that make amputation inevitable (Rutherford Category 6)
* Active clinical infection within one week of enrollment
* Treatment with immunosuppressant drugs
* Known drug or alcohol dependence, or any other factors which will interfere with the study conduct or interpretation of the results
* Not suitable to participate in the opinion of the principal investigator
* History cancer (other than non-melanoma skin cancer or in situ cervical cancer) within five years preceding study entry
* Unwilling and/or not able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Improvement from baseline in perfusion as measured by ankle-brachial index and collateral artery number | 6 months
  Contrast Angiography
Number of adverse events reported | 6 months

SECONDARY OUTCOMES:
Improvement from baseline in improvement or resolution of ulcer or gangrene | 3 months, 6 months
  Visual assessment
Limb Salvage | 3 months and 6 months
  Assessed with doppler to measure blood flow to the affected area.

OTHER OUTCOMES:
Change from baseline in Quality of Life | 3 months, 6 months
  King's College Hospital's Vascular Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided